CLINICAL TRIAL: NCT05230108
Title: Implementation of Advanced Triage in the Emergency Department of Bellvitge University Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Official Barcelona Nurses Association (COIB) (Unknown)
Responsible Party: Principal Investigator, Cristina Font Cabrera, Emergency Nurse, Hospital Universitari de Bellvitge
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PR085/20
Record Dates: First submitted 2021-12-22; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Nurse's Scope of Practice
Keywords: advanced practice nurse emergency; Advanced Interventions Nursing; Emergency Department.
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: The fourth step is a quasi-experimental study consisting of two phases: the first, a retrospective control phase, and the second, a prospective intervention phase in which advanced triage will be implemented. In phase 1, control, quality of care indicators will be assessed, based on quality indicators in the emergency department, waiting time and satisfaction, and the level of pain. In addition, different epidemiological, socio-cultural and clinical variables will be measured. In phase 2, the intervention phase, advanced triage will be implemented based on advanced practices nurse and the indicators of quality of care and pain will be assessed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 (F1): retrospective control. (No Intervention): Phase 1, retrospective, will include all patients who attended the ED from January 2018 to December 2022.
- Phase (F2): prospective intervention of Advanced Triage (Experimental): Phase 2, prospective, where advanced triage based on advanced practice nurse will be implemented. Will include patients from January 2023 to December 2024.
  Interventions: Procedure: Advanced Triage

INTERVENTIONS:
Procedure: Advanced Triage — Advanced triage is an intervention that allows the emergency nurse to resolve health problems of low clinical complexity. All actions are aimed at resolving a health problem based on a protocol previously agreed upon by a multidisciplinary team.
  Other Names: Advanced triage is part of advanced practice nurse (APN).
  Arms: Phase (F2): prospective intervention of Advanced Triage

SUMMARY:
This study evaluates the efficacy of advanced triage in improving the quality of care outcomes of patients attending the Emergency Department (ED) united care of high complexity hospital.

There are four steps; Step 1 will consist of a concept analysis. Step 2 will include a mapping of advanced practice protocol terminologies. Step 3 will analyse the opinion of health professionals on advanced triage. In step 4: in retrospective phase, sociodemographic and clinical variables and quality indicators such as waiting time will be analysed. After that, in the prospective phase, advanced triage will be implemented and the two cohorts will be compared.

DETAILED DESCRIPTION:
STEP 1:

Study design: a concept analysis will be carried out based on a systematic analysis method by which it details and specifies the element to be studied, in this case, the Advanced Triage (AT). This study is based on the method that was outlined by Wilson (Wilson, 1969) and later evolved by Avant (Walker & Avant, 1989). This technique consists of eleven stages: 1) isolating questions concerning the concept; 2) finding suitable answers; 3-7) developing real or invented cases; 8) determining the social context; 9) identifying the underlying emotions; 10) establishing the practical results; 11) defining the results in language that facilitates the clarification of the controversial concept. The use of this methodology provides the construction of different definitions that reach all variants of the AT concept.

STEP 2:

Study design: Observational, descriptive, cross-sectional, retrospective, retrospective, observational study of interobserver concordance of bidirectional cross-mapping between Architecture Terminology Interface Knowledge (ATIC), Nursing Diagnoses: Definitions & Classification (NANDA), Nursing Interventions Classification (NIC) and the International Classification of Diseases and Related Health Problems (ICD-10). Based on the protocols of the Nurse Demand Management (NDM) for primary health care (PHC) of the Catalan Institute of Health.

Data collection: The data collector will proceed to design a form that allows the collection and connection of the three terminologies in each concept (assessment, diagnosis and intervention). The identification of these equivalences will be carried out by the participation of three nurses independently of each of the researchers. Several interobserver consensus sessions will be held according to the results of the concordance. Discrepancies will be resolved, if appropriate, through the agreement processes. To make the equivalences of the concepts included in the NDM protocols with the different languages (ATIC, NANDA, NIC and ICD-10), with trichotomous variables: Yes /No/ Partially; and nominal quantitative variables, to facilitate the understanding of the mapping, the codes representing the type of equivalence are included.

Data analysis: The collected data will be processed and checked for processing errors and analysed with EXCEL. Interobserver reliability will be calculated by considering the ratio according to the results of the three investigators and using the kappa(K) index calculation, in which the agreement is considered to be: (1) low, if (k) ≤0.20; (2) moderate, if (k) 0.21-0.40; (3) acceptable, if (K) 0.61-0.80 and (5) excellent, if (k) ≤0.81.

STEP 3 Study design: observational, descriptive, cross-sectional and prospective study of the different protocols already existing in the PHC of the Catalan Institute of Health and assess whether they are suitable for the hospital setting

Study setting: The study will be carried out in the ED of a high complexity public hospital in the southern metropolitan area of Barcelona (Spain). This stage will consist of two phases:

Phase 1 (P1): a committee of experts will be formed, which will evaluate the existing protocols. Phase 2 (P2): surveys will be passed to several health professionals working in the ED of a high complexity hospital, in order to know their opinion about the AT.

Participants: In Phase 1, it will consist of 12 healthcare professionals (8 nurses and 4 doctors) who will work in the ED of a high complexity hospital. In Phase 2, the study population will be all healthcare professionals who work in the ED in an assisting or management capacity in a high complexity hospital.

Selection criteria:

Inclusion criteria: nurses and physicians, assistants and managers of the emergency departments of public hospitals in Catalonia.

Exclusion criteria: Auxiliary nursing care technicians, orderlies, nurses and administrative staff.

Sample size (phase 2):Starting from a maximum indeterminacy with an expected proportion (p)= 0.05, a 95% confidence interval (α=0.05) and a precision (y)=0.05. The number of professionals to be included will be 385. Assuming 15% of possible losses, the corrected sample formula will be applied, which gives a total sample of 490 individuals. The sampling technique in this phase will be non-probabilistic consecutive sampling.

Data collection: the variables for phase 1 and phase 2 of stpe 3 will be the usefulness and applicability of the NDM, protocols by the hospital AT and two lines will be considered: the first, the evaluation of the perception of usefulness and the second, of applicability by the healthcare professionals, from the two phases.

Perception of usefulness: (phases 1 and phases 2) professionals' impression and assessment of the correctness and advantages of each of the 33 protocols of the NDM by the AT. This variable is measured on a qualitative ordinal scale: 0 to 10, where 0 feels totally disagree and 10 feels totally agree.

Perception of applicability: (phases 1 and phases 2) practitioners' impression and assessment of the adaptability and feasibility of each of the 33 NDM protocols by AT. This variable is measured with an ordinal qualitative scale: 0 to 10, feeling 0 strongly disagree and 10 strongly agree.

Secondary variables: (phases 2) years of experience, professional groups, beliefs about nursing professional domains, knowledge about AT and opinion about AT.

The data collection in phase 1 will be carried out on the basis of grids, where the 33 protocols of the NDM will be analysed. In each protocol, 12 questions will have to be analysed. In phase 2, a questionnaire consisting of four blocks will be administered: (1) socio-demographic data will be asked; (2) knowledge of the AT will be asked; (3) the opinion held by the different health professionals will be asked; (4) nursing competences will be asked.

Data analysis: qualitative variables will be described by proportions, calculating 95% confidence intervals. Quantitative variables will be described with mean and median as measures of centrality, and standard deviation and interquartile range as measures of dispersion.The normality of the distribution of the quantitative variables will be checked with the Kolmogorov-Smirnov test pot, and the parametric and non-parametric pots indicated in each case in the bivariate analysis will be applied; normally, the most commonly used pots will be the Chi-square, the Mann-Whitney U, the Student's t and Pearson's correlation-regression pots. Finally, multivariate analysis will include logistic regression techniques. P-values of less than 0.05 will be considered statistically significant.

STEP 4:

Study design: quasi-experimental study consisting of 2 phases: phase 1 (retrospective control) and phase 2 (prospective intervention), where the AT will be implemented based on the advanced nurse practitioner's.

Study setting: the scope of the study will be the ED of a highly complex hospital in a centre in Catalonia (northeastern Spain), which serves as a community reference for 201,192 inhabitants of Hospitalet and Prat de Llobregat and is a reference centre for processes requiring high technology for more than 2 million inhabitants of the South Metropolitan area, Camp de Tarragona and Terres de l'Ebre. Outpatient ED of a tertiary-care centre in Catalonia (Northeast Spain), which serves as a referral centre for community reference of 201,192 people in the Southern Metropolitan Area of Barcelona.

In both phases, all adult patients (>18 years) who will visit the hospital ED and who will be classified with priority levels III, IV or V on the Emergency Severity Index (ESI) scale will be eligible to participate in the study.

Procedure and interventions:

Control group will apply the usual care of the service and will be analysed: (a) quality indicators specific to triage; (b) cluster; (c) satisfaction; (c) pain; (d) waiting time. This part of the study will allow us to gain a better understanding of the reality of ED care. In relation to the level of urgency and its complexity, allowing us to establish the digital footprint. In order to be able to compare them with each other.

Data analysis: qualitative variables will be described by proportions, calculating 95% confidence intervals. Quantitative variables will be described with mean and median as measures of centrality, and standard deviation and interquartile range as measures of dispersion. The normality of the distribution of quantitative variables will be checked with the Kolmogorov-Smirnov test, and the parametric and non-parametric pots indicated in each case in the bivariate analysis will be applied; normally, the most commonly used pots will be the Chi-square, the Mann-Whitney U, the Student's t and Pearson's correlation-regression pots. Finally, multivariate analysis will include logistic regression techniques. P-values of less than 0.05 will be considered statistically significant. All data will be analysed using Statistical Package for the Social Sciences (SPSS) v26.0 software.

The final results will be used to design the hospital ED TA implementation programme.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age, admitted to EDs classified with Emergency Severity Index (ESI) severity levels III, IV and V.

Exclusion Criteria:

* patients over 70 years of age
* pregnant women
* patients with a Glasgow Glasgow score of less than 15
* patients with more than 3 chronic pathologies and/or 1 complex chronic
* disease or patients reconsulting the ED for the same reason for consultation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality indicators specific to triage. | Pre-intervention time as an initial reference.
  Set of peculiar traits that characterise someone or something. This variable is a composite variable which is made up of quality indicators specific to triage, waiting time, and variables to inform the sample.
  * Arrival/registration-triage time: The time from patient arrival at the ED to triage classification. Quality indicators define this time as <= 10 minutes (min) over the total number of patients triaged.
  * Waiting time to be visited: It is established that at least 90% of patients must be visited by a medical team within <= 120 min from their classification, and 100% within <= 240 min

SECONDARY OUTCOMES:
Cluster: | Throgh study completion, an average of 1 year.
  This variable allows grouping several individuals in similar conditions. This variable is composed of:
  * Age (18-75 years)
  * Sex: Male/Female
  * Country of origin: Patient birth country.
  * Origin of the patient: Indicates whether a patient arrives at the emergency department referred from another health resource or not. The following values are coded: (a) home (b) residence, (c) primary care, (d) hospital, (e) hospitalisation at home, (f) other outpatient care.
CatSalut-PLAENSA© | 12 months.
  This scale allows us to measure the satisfaction of patients who will be seen in the ED. The CatSalut-PLAENSA© satisfaction survey is based on an ordinal scale from 0 to 10. This variable will be measured on a qualitative ordinal scale; from 0 to 10, with 0 being totally disagree and 10 being totally agree.
Waiting times | 12 months.
  This will be analysed using the hospital's computer system. The following will be recorded: time of entry to the ED, time of triage, time of attendance (nurse or doctor), time of administration of analgesia, time of discharge from the ED and total time the patient has been in the emergency department.
The Visual Analog Scale (VAS or EVA) | 12 months.
  is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." This variable is measured on an ordinal qualitative scale; 0 to 10, with 0 being no pain and 10 being very intense pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Austin EE, Blakely B, Tufanaru C, Selwood A, Braithwaite J, Clay-Williams R. Strategies to measure and improve emergency department performance: a scoping review. Scand J Trauma Resusc Emerg Med. 2020 Jun 15;28(1):55. doi: 10.1186/s13049-020-00749-2. PMID 32539739
- [Background] Bittencourt RJ, Stevanato AM, Braganca CTNM, Gottems LBD, O'Dwyer G. Interventions in overcrowding of emergency departments: an overview of systematic reviews. Rev Saude Publica. 2020;54:66. doi: 10.11606/s1518-8787.2020054002342. Epub 2020 Jul 3. PMID 32638885
- [Background] Butti L, Bierti O, Lanfrit R, Bertolini R, Chittaro S, Delli Compagni S, Del Russo D, Mancusi RL, Pertoldi F. Evaluation of the effectiveness and efficiency of the triage emergency department nursing protocol for the management of pain. J Pain Res. 2017 Oct 16;10:2479-2488. doi: 10.2147/JPR.S138850. eCollection 2017. PMID 29081670
- [Background] Hinson JS, Martinez DA, Schmitz PSK, Toerper M, Radu D, Scheulen J, Stewart de Ramirez SA, Levin S. Accuracy of emergency department triage using the Emergency Severity Index and independent predictors of under-triage and over-triage in Brazil: a retrospective cohort analysis. Int J Emerg Med. 2018 Jan 15;11(1):3. doi: 10.1186/s12245-017-0161-8. PMID 29335793
- [Background] Innes K, Jackson D, Plummer V, Elliott D. Emergency department waiting room nurse role: A key informant perspective. Australas Emerg Nurs J. 2017 Feb;20(1):6-11. doi: 10.1016/j.aenj.2016.12.002. Epub 2017 Jan 17. PMID 28108139
- [Background] Lauks J, Mramor B, Baumgartl K, Maier H, Nickel CH, Bingisser R. Medical Team Evaluation: Effect on Emergency Department Waiting Time and Length of Stay. PLoS One. 2016 Apr 22;11(4):e0154372. doi: 10.1371/journal.pone.0154372. eCollection 2016. PMID 27104911
- [Background] Sarria-Guerrero JA, Luaces-Cubells C, Jimenez-Fabrega FX, Villamor-Ordozgoiti A, Isla Pera P, Guix-Comellas EM. Pediatric televisits and telephone triage: impact on use of a hospital emergency department. Emergencias. 2019 Ago;31(4):257-260. English, Spanish. PMID 31347806
- [Background] Woo BFY, Lee JXY, Tam WWS. The impact of the advanced practice nursing role on quality of care, clinical outcomes, patient satisfaction, and cost in the emergency and critical care settings: a systematic review. Hum Resour Health. 2017 Sep 11;15(1):63. doi: 10.1186/s12960-017-0237-9. PMID 28893270
- [Background] Zachariasse JM, van der Hagen V, Seiger N, Mackway-Jones K, van Veen M, Moll HA. Performance of triage systems in emergency care: a systematic review and meta-analysis. BMJ Open. 2019 May 28;9(5):e026471. doi: 10.1136/bmjopen-2018-026471. PMID 31142524
- [Derived] Font-Cabrera C, Juve-Udina ME, Galimany-Masclans J, Fabrellas N, Rosello-Novella A, Sancho-Agredano R, Adamuz J, Guix-Comellas EM. Implementation of advanced triage in the Emergency Department of high complexity public hospital: Research protocol. Nurs Open. 2023 Jun;10(6):4101-4110. doi: 10.1002/nop2.1622. Epub 2023 Jan 31. PMID 36719704